CLINICAL TRIAL: NCT07373171
Title: Evaluation of Different Sizes of Left-Sided Double-Lumen Tubes for Thoracic Surgery in a Tertiary Level Teaching Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Jog Adhikari, MD resident Doctor, Tribhuvan University, Nepal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 258/0821083
Record Dates: First submitted 2025-12-18; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Lung Adenocarcinoma; Lung Abscess
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Abscess

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 35 Fr group (Experimental)
  Interventions: Device: Intubation of patients undergoing thoracic surgery with left sided double lumen tube
- DLT size according to height (No Intervention)

INTERVENTIONS:
Device: Intubation of patients undergoing thoracic surgery with left sided double lumen tube — During the intervention Integrity of the tracheal and bronchial cuffs will be checked first. Lubrication of the outside of the 35 Fr DLT will be done using 2.5% lidocaine jelly and intubating stylet will be inserted (can be preshaped to aid placement of the DLT). Direct laryngoscopy will be done to visualize the glottis. DLT will be advanced till the endobronchial cuff is passed beyond the vocal cords and then the stylet is removed. DLT will be rotated 90 anticlockwise and the tracheal cuff is inserted beyond the glottis until resistance is encountered.
  Arms: 35 Fr group

SUMMARY:
Double lumen tubes (DLT) have become standard of care for one lung ventilation in thoracic and esophageal surgeries. Selection of accurate size of DLT is important to achieve proper one lung ventilation, prevent trauma to airway, easy intubation, prevention of displacement of DLT and adequate oxygenation intraoperatively. There are no definitive guidelines to select the correct size of DLT. The aim of this study is to observe if there is any difference in the number of intubation attempts, intraoperative oxygenation and postoperative sore throat while using 35 Fr DLT size and other DLT size. The research will be conducted between Ashoj 1st 2082 to Chaitra 30 2082 at Manmohan Cardiothoracic Vascular and Transplant Center(MCVTC). Fifty patients aged more than eighteen years undergoing thoracic surgery requiring One Lung Ventilation(OLV) with left sided DLT will be selected for the study. Participants will be randomly assigned to 35 Fr DLT size group or DLT size group according to the height. Patients in both the groups will be given the samepreoperative care, intraoperative care and postoperative care. Besides patient's demography, diagnosis and operative procedure; number of intubation attempts, modified Cromack-Lehane(CL) grade, size of DLT, intraoperative oxygen saturation SpO₂ and postoperative sore throat on day of surgery and first postoperative day will be recorded. Statistical analysis will be done using t- test for independent variable, confidence interval for outcome of sore throat, significance of difference for number of male and female; rates, risk ratio and odds ratio will be calculated using 2x2 contingency table. P ≤ 0.05 will be considered statistically significant. Our expected outcome is 35 Fr DLT are easier to intubate, does not affect intraoperative oxygenation and decrease the incidence of postoperative sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older undergoing thoracic surgery requiring OLV with placement of a left-sided DLT

Exclusion Criteria:

* Patient refusal
* Need for rapid sequence intubation (RSI) due to increased aspiration risk
* Anticipated difficult intubation
* Emergency surgery
* Patient already intubated with a single-lumen ET tube
* DLT tube change to single lumen tube at the end and shifted with ETT in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Ease of intubation using a 35 Fr DLT | Day 1
  Ease of intubation is assessed using "number of intubation attempt and "Cormack-Lehane grade" that will be determined by anaesthesia provider who is intubating. The number of intubation attempt is the tube pass attempt during intubation and Cormack-Lehane grade is the percentage of vocal cord structure visualized during direct laryngoscopy. Number of intubation attempt and cormack-Lehane grading will be recorded in the proforma of the study.
Difference in intraoperative oxygenation between 35 Fr and different sizes of DLT | Day 1
  The percentage of oxygen saturation( SpO2 %) will be recorded at 5 minutes and 10 minutes after one lung ventilation from the ventilator monitor attached to the patient in the operation room. The percentage of oxygen saturation will be recorded in the study proforma and later compared between the groups.
Postoperative sore throat | Day 2
  Postoperative sore throat will be assessed using a yes/no question asked by an attending nurse in the post operative ward within 24 hours of postoperative period. If the patient has sore throat then it will be graded.
  The question and grade will be as follow Do you have a sore throat: (yes/no) if the answer is yes then graded as 0 = no sore throat
  1. = mild sore throat (complains of sore throat only on asking)
  2. = moderate sore throat (complains of sore throat on his/her own) 3= severe sore throat (change of voice or hoarseness, associated with throat pain The answer and grade will be recorded and later analysed between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Manmohan Cardiothoracic Vascular and Transplant Centre, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Allocated group of participant, participant demographic, primary and secondary outcomes, data analysis and result will be shared after completion of the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be shared after completion of the study and will be available for 12 months.